CLINICAL TRIAL: NCT06883851
Title: Evaluating the Efficacy of Structured Pelvic Floor Muscle Rehabilitation Combined With Desmopressin in the Management of Primary Monosymptomatic Nocturnal Enuresis in Children
Brief Title: Effectiveness of Pelvic Floor Muscle Rehabilitation Combined With Desmopressin in Children With Primary Monosymptomatic Nocturnal Enuresis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Private Selcuk Sılay Pediatric Urology Clinic (Unknown); Medipol Acıbadem Regional Hospital (Unknown)
Responsible Party: Principal Investigator, Aygul Koseoglu Kurt, Principal investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-6971
Record Dates: First submitted 2025-03-11; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Primary Nocturnal Enuresis; Nocturnal Enuresis in Children
Keywords: biofeedback; core stabilization; exercise; urinary incontinence; management; treatment; enuresis; pelvic floor rehabilitation; desmopressin
MeSH Terms: conditions — Motor Activity; Urinary Incontinence; Enuresis

STUDY DESIGN:
Intervention Model Description: Children aged 7 to 13 years, diagnosed with PMNE and meeting the inclusion criteria, will be included in the study. The sample size for the study will be determined after data collection from a pilot study involving ten participants.
Masking Description: The children included in the study will be randomized into two groups: the control group (CG) and the Structured Pelvic Floor Muscle Rehabilitation Group (SPFMRG), following the completion of evaluations by the pediatric urologist. The participants will be randomly assigned to groups using the website https://www.randomizer.org/.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (No Intervention): The group that will receive first-line treatment, consisting of classic DDVAP treatment with evidence level A and urotherapy training, will be included in the treatment of PMNE. The DDVAP dosage will be determined and prescribed by the pediatric urologist. Only these treatments will be applied, and no pelvic floor rehabilitation will be implemented.
- Structered Pelvic Floor Muscle Rehabilitation Group (SPFMRG) (Experimental): This group will receive, in addition to the DDVAP therapy prescribed by the pediatric urologist and urotherapy training, 10 weeks of structured pelvic floor muscle rehabilitation sessions.
  Interventions: Other: Structured pelvic floor rehabilitation

INTERVENTIONS:
Other: Structured pelvic floor rehabilitation — The classic DDVAP therapy will be administered by the pediatric urologist. The classic urotherapy training recommended for enuresis will be provided by the physiotherapist. In addition, structured pelvic floor muscle rehabilitation (SPFMR) will be provided by the physiotherapist for 10 weeks. Each session is planned to last approximately 60 minutes.
  SPFMR will include multiple interventions combined. Below is information about the brief interventions.
  * Diaphragmatic Breathing Training
  * Pelvic Floor Training with Biofeedback
  * Core Stabilization Exercises
  * Squat Exercises
  * External Rotator Strengthing
  * Adductor Strengthing
  * Balance Training
  * Home Exercises
  Arms: Structered Pelvic Floor Muscle Rehabilitation Group (SPFMRG)

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effects of Structured Pelvic Floor Muscle Rehabilitation (SPFMR) in children with Primary Monosymptomatic Nocturnal Enuresis (PMNE) who are undergoing desmopressin asetat (DDAVP) treatment prescribed by a pediatric urologist. The study aims to investigate whether SPFMR can reduce the frequency and severity of enuresis episodes and whether it can also reduce relapse rates in the short- and long-term follow-up. The main questions the study seeks to answer are:

* Does SPFMR reduce the frequency and severity of enuresis episodes in children with PMNE?
* Does SPFMR treatment reduce relapse rates in children with PMNE in the long term? Researchers will compare the group receiving SPFMR in addition to DDAVP treatment with a control group receiving only DDAVP treatment. This comparison will help evaluate the effect of SPFMR on the severity of enuresis episodes and relapse rates.

Participants will:

* Receive DDAVP treatment (SPFMR group and Control group)
* Participate in SPFMR sessions ( SPFMR group)
* Keep a diary of enuresis frequency and severity
* Assess relapse during short- and long-term follow-up

The hypotheses of the study are:

H0: Adding SPFMR to desmopressin treatment for children with PMNE has no short-term effect on the severity of enuresis episodes.

H1: Adding SPFMR to desmopressin treatment for children with PMNE has a short-term effect on the severity of enuresis episodes.

H0: Adding SPFMR to desmopressin treatment for children with PMNE has no long-term effect on the severity of enuresis episodes.

H2: Adding SPFMR to desmopressin treatment for children with PMNE has a long-term effect on the severity of enuresis episodes.

DETAILED DESCRIPTION:
Nocturnal enuresis (NE) is defined as nighttime urinary incontinence (bedwetting) during sleep in a healthy child older than five years, occurring at least twice a week for at least three consecutive months, sufficient to wet most or all of the sleeping area. NE is categorized into two types based on the presence or absence of daytime lower urinary tract symptoms (LUTS): monosymptomatic nocturnal enuresis (MNE) and non-monosymptomatic nocturnal enuresis (NMNE). MNE refers to involuntary nighttime urinary incontinence during sleep in children older than five years without any congenital or acquired urological or central nervous system (CNS) disorders and without daytime LUTS.

Approximately 80% of children diagnosed with NE are classified as having MNE. NE is further subdivided into primary and secondary subgroups based on the onset period. Primary NE refers to children who have had less than six months of dryness since toilet training, whereas secondary NE is diagnosed in children who have experienced six months or more of dryness since toilet training . In summary, primary MNE is used to diagnose children who have had less than six months of nighttime dryness since toilet training and lack daytime LUTS.

NE, previously viewed as a psychiatric disorder, is now understood to involve a variety of mechanisms and multifactorial causes. Studies suggest that children with NE exhibit a range of symptoms across different systems. The current understanding of NE's etiology includes three main factors:reduced noctural bladder capacity, nocturnal polyuria and decreased arousability during sleep.

Treatment options for MNE include urotherapy (healthy bladder and bowel training), enuresis alarms (bedwetting alarms), and pharmacological agents such as desmopressin acetate (DDAVP), anticholinergics, and tricyclic antidepressants. These methods can be used alone or in combination for the treatment of MNE. Among first-line treatments, enuresis alarms (evidence level 1A) and DDAVP (evidence level 1A) are widely accepted approaches in pediatric urology. It is estimated that approximately one-third of enuretic children may require additional treatment following first-line interventions.

DDAVP is a pharmacological agent developed as an analog of vasopressin or antidiuretic hormone. Its antienuretic effect reduces the volume of urine produced overnight, allowing the bladder to store the produced urine. Literature reports that about one-third of children undergoing DDAVP therapy achieve reliable dryness while on the medication, another third experience moderate benefits, and the remaining third see no benefit Although high relapse rates of NE have been reported following the cessation of DDAVP treatment, a recent meta-analysis showed that structured dose-dependent discontinuation of DDAVP provides better relapse-free rates.

Although DDAVP and alarm therapy, both with evidence level 1A, are established first-line treatments for MNE, research continues into additional therapies and complementary approaches that may enhance treatment success. These include chiropractic therapy, homeopathy, pelvic floor exercises, electrotherapy, breathing exercises, hypnosis, Ayurveda, reflexology, traditional Chinese and Iranian medicine, massage, yoga, and herbal treatments.

Considering the potential pharmacological side effects and the lack of adherence among families, DDAVP alone may be insufficient for treating PMNE. Additionally, given the deviations in pelvic floor muscle (PFM) activation values reported in enuretic children, it is necessary to investigate a combined approach incorporating PFM rehabilitation into medical treatment for children diagnosed with PMNE. The study's hypothesize is Structured Pelvic Floor Muscle Rehabilitation (SPFMR), applied to children with PMNE who are already receiving DDAVP therapy (as prescribed by a pediatric urology physician), will reduce the frequency and severity of enuresis episodes and decrease relapse rates in both short- and long-term follow-ups.

The study protocol will adhere to applicable regulations, the current Declaration of Helsinki, and the principles of Good Clinical Practice. Since participants are under the age of 18, written and verbal consent will be obtained from their parents. The study will commence after receiving ethics committee approval and completing the clinical trial registration.

Physiotherapy Modalities to Be Used in Structured Pelvic Floor Muscle Rehabilitation (SPFMR):

- Diaphragmatic Breathing Training: The diaphragm is not only a respiratory muscle but also a part of the core system. It works synergistically with PFM to ensure the proper function of the pelvic floor. ]. The diaphragm plays a vital role in generating proper intra-abdominal pressure and transmitting it from the cranial to the caudal regions. Additionally, the pushing pressure generated by the diaphragm is crucial for voiding (urination, defecation, and childbirth) and the functional activity of PFM. In PFMRG, diaphragmatic breathing exercises will involve inhaling through the nose for 4 seconds and exhaling through the mouth for 8 seconds in a series of 30 repetitions lasting approximately 6 minutes. Breaks will be given in case of dizziness or discomfort, after which the exercises will resume.

- Biofeedback-Assisted PFM Training Biofeedback therapy is a non-invasive, easily accessible technique for treating pediatric pelvic floor dysfunction. As a physical therapy modality, biofeedback aims to train appropriate PFM activity essential for normal, healthy bowel and bladder function. Electromyographic biofeedback is the most commonly used type for treating these dysfunctions. Biofeedback therapy is an instrument-based learning process that uses operant conditioning. It provides visual, auditory, and verbal feedback to promote self-control over physiological processes that are otherwise outside awareness or under limited voluntary control, such as autonomic and neuromuscular activity.

Before starting each session, the microvolt value produced by submaximal muscle contraction will be measured three times and recorded using the Libert Phenix device. The CE certificate and registration of the device with the Ministry of Health are provided. Subsequently, PFM will be trained with 15-second phasic contractions at 30%, 60%, and 90% of submaximal strength, followed by 10 seconds of relaxation to achieve basal relaxation. Each phasic contraction training period will be completed in 25 seconds. The phasic training period will include 24 repetitions completed in 600 seconds (10 minutes).

Following phasic contraction training, tonic contraction exercises will be performed at 30% muscle contraction based on recorded submaximal activation. Each tonic contraction will last for 10 seconds, followed by a 10-second relaxation period to achieve basal relaxation, with one tonic contraction cycle completed in 20 seconds. The tonic contraction training period will consist of 30 repetitions, completed in 600 seconds (10 minutes). The endurance training, starting at 30%, will gradually progress to 40%, 50%, 60%, and 80%.

SPFMRG participants will be taught to perform proper PFM contractions without engaging their adductor or gluteal muscles. Training will begin in the supine position and progress to seated and then standing positions to introduce gravitational effects over the weeks.

- Core Stabilization and Combined Squat Exercises: In addition to ensuring continence and supporting various pelvic organs, PFMs are a component of the local stabilization system, playing a critical role in the lumbopelvic region in association with the transversus abdominis and multifidus muscles. These muscles work synergistically with other muscles surrounding the abdominal cavity, such as the anterolateral abdominal muscles and thoracic diaphragm, to regulate intra-abdominal pressure and ensure abdominal stability. Core stabilization exercises will follow the Dynamic Neuromuscular Stabilization (DNS) method, based on developmental kinesiology. DNS focuses on the integrated spinal stabilization system, targeting deep cervical flexors, the diaphragm, transversus abdominis, multifidus, and PFMs, by mimicking stabilization patterns observed in healthy infants.

DNS exercises aim to activate the spinal stabilization system effectively through repetition and help individuals regain control during various tasks. While DNS methods have been studied for urinary incontinence in adults, studies are needed on pediatric incontinence. DNS methods have been applied in pediatric populations with cerebral palsy.

DNS Exercises:

* Crawling Bug: Supine position with a 55 cm Pilates ball positioned between the feet and hands, rotating the ball 5 times x 3 sets.
* Rocking Bear: Quadruped position, lifting and lowering the knees 5 cm above the mat, 10 repetitions x 3 sets.
* Reaching Cat: Cross-extension exercise with a resistance band looped around the foot, one end held by the participant in a quadruped position, 10 repetitions x 3 sets.
* Showering Elephant: Holding a 55 cm Pilates ball between the hands, synchronizing squats with lifting the ball to shoulder height, 10 repetitions x 3 sets.
* External Rotator and Adductor Strengthening:

Strengthening the external rotator muscles, including the obturator internus (OI), has been shown to play a synergistic role in enhancing PFM function and strength. It has also been reported as an easily applicable and comprehensible auxiliary exercise for women with reduced PFM contraction ability. While studies on the role of OI in PFM rehabilitation are abundant in adult women, pediatric studies are limited and primarily case studies . Participants will perform abduction and external rotation of the lower extremities with a resistance band placed between the knees, 10 repetitions x 3 set.

While studies on the role of OI in PFM rehabilitation are abundant in adult women, pediatric studies are limited and primarily case studies. Participants will perform abduction and external rotation of the lower extremities with a resistance band placed between the knees, 10 repetitions x 3 set.

- Balance Training: Participants will perform balance exercises on a Bosu ball in both double-leg and single-leg stances, with eyes open and closed, for 30 seconds x 3 sets.

- Home Exercises: Participants will be asked to perform the following home exercises three times per week.

* Diaphragmatic breathing exercises: Inhaling for 4 seconds, exhaling for 8 seconds, 30 repetitions (approximately 6 minutes).
* PFM contractions: 10 seconds of contraction, followed by 10 seconds of relaxation, for 6 cycles.
* 10 squat exercises.
* Crawling Bug and Rocking Bear exercises: 30 seconds x 3 sets. Participants will be provided with a home exercise tracking chart, monitored weekly by the research physiotherapist.

After the treatment, participants' dry nights and symptoms will be converted into percentages following the ICCS treatment outcome recommendations. According to this recommendation, a reduction of less than 50% in symptoms will be considered no response to treatment; a reduction of 50% to 99% in symptoms will be considered a partial response, and the complete resolution of symptoms (100% reduction) will be considered full success.

ELIGIBILITY:
Inclusion Criteria:

* Being between 7 and 13 years old
* Diagnosed with primary MNE by a pediatric urology department within the last 6 months
* No urinary tract infection verified by laboratory tests
* Ability to communicate in Turkish and absence of mental deficit
* No diagnosed psychiatric problems
* Willingness to participate in the study (child and family)

Exclusion Criteria:

* Presence of orthopedic conditions preventing evaluation
* Anatomical anomalies in the urinary system
* History of urinary system surgery
* Neurological disorders
* Presence of mental retardation
* History of orthopedic surgery that could alter pelvic or lower extremity integrity
* Receiving PFM rehabilitation in the last 6 months
* Using nighttime alarm therapy in the last 6 months
* Receiving any treatment for enuresis in the last 6 months

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-03-11 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
The Nighttime Bedwetting Diary | baseline; 10th week after baseline; 12th week after baseline and 16th week after baseline
  The diary records dry and wet nights, the amount of bedwetting, bedtime, and wake-up time. The nighttime bedwetting diary will be completed one week before treatment initiation, during the treatment period (10 weeks), and throughout the follow-up phase for both groups. Data will be shared weekly with the researchers, either face-to-face or via phone (WhatsApp, email, etc.).

SECONDARY OUTCOMES:
Uroflowmetry Test | baseline; 10th week after baseline; 12th week after baseline and 16th week after baseline
  During the uroflowmetry evaluation, patients will be asked to urinate into a sensor-equipped uroflowmetry container (MMES ® brand) when they feel the urge to urinate. For children whose feet do not touch the ground, a stool will be used to ensure a proper toilet position. To minimize external factors affecting the urination pattern, it will be ensured that no one else is present in the uroflowmetry room except the patient. The parameters obtained from the measurement will be used to evaluate the voiding phase of the bladder. Flow rate will be recorded. Flow rate is the volume of urine per unit of time, typically expressed in milliliters per second (ml/s).
Post-Void Residual (PVR) Assessment | baseline; 10th week after baseline; 12th week after baseline and 16th week after baseline
  The Clarius® transabdominal ultrasound device will be used, and measurements will be performed from the suprapubic region. During the measurement, the patient will be positioned in a supine position with knees slightly flexed and supported with a towel beneath. The volume values calculated by the probe in the coronal and sagittal regions in mm³ will be automatically multiplied by the ultrasound system to calculate the residual urine volume in the bladder.
Bladder Diary | baseline; 10th week after baseline; 12th week after baseline and 16th week after baseline
  The diary will be maintained over a 48-hour period, recording daytime voiding frequency, voided volume, fluid types, and the amounts.
Pelvic Floor Muscle Activation Measurement | baseline; 10th week after baseline; 12th week after baseline and 16th week after baseline
  After proper placement of the electrodes, PFM activity will be measured using the NeuroTrac Myoplus4 Pro device. The CE certificate and registration of the device with the Ministry of Health are presented. Participants will be asked to perform 5 seconds of maximal contractions of their PFM ("work" phase EMG activity) followed by 5 seconds of relaxation ("rest" phase EMG activity), repeated in succession after resting. The device provides verbal commands of "work" for each contraction and "rest" for each relaxation. The measurement lasts for 55 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Pisirici, Assist. Prof., Study Director — Bahçeşehir University; Mesrur Selcuk Silay, Prof. Dr., Study Chair — Medipol University; Aygul Koseoglu Kurt, Ph.D. (c), Principal Investigator — Bahçeşehir University
Locations (2):
- Turkey (Türkiye) (2):
  - Private Selcuk Silay Pediatric Urology Clinic, Istanbul, Beşiktaş
  - Medipol Acıbadem Region Hospital, Istanbul, Kadıkoy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reilly M, Homsy Y. Treatment of a child with daytime urinary incontinence. Pediatr Phys Ther. 2008 Summer;20(2):185-93. doi: 10.1097/PEP.0b013e318171fb8d. PMID 18480719
- [Result] Kim DH, An DH, Yoo WG. Effects of 4 weeks of dynamic neuromuscular stabilization training on balance and gait performance in an adolescent with spastic hemiparetic cerebral palsy. J Phys Ther Sci. 2017 Oct;29(10):1881-1882. doi: 10.1589/jpts.29.1881. Epub 2017 Oct 21. PMID 29184312
- [Result] Bo K. Pelvic floor muscle training is effective in treatment of female stress urinary incontinence, but how does it work? Int Urogynecol J Pelvic Floor Dysfunct. 2004 Mar-Apr;15(2):76-84. doi: 10.1007/s00192-004-1125-0. Epub 2004 Jan 24. PMID 15014933
- [Result] Ladi-Seyedian SS, Sharifi-Rad L, Nabavizadeh B, Kajbafzadeh AM. Traditional Biofeedback vs. Pelvic Floor Physical Therapy-Is One Clearly Superior? Curr Urol Rep. 2019 May 30;20(7):38. doi: 10.1007/s11934-019-0901-9. PMID 31147796
- [Result] Wagner B, Steiner M, Huber DFX, Crevenna R. The effect of biofeedback interventions on pain, overall symptoms, quality of life and physiological parameters in patients with pelvic pain : A systematic review. Wien Klin Wochenschr. 2022 Jan;134(Suppl 1):11-48. doi: 10.1007/s00508-021-01827-w. Epub 2021 Mar 22. PMID 33751183
- [Result] Hodges, P., R. Sapsford, and H. Pengel, Feedforward activity of the pelvic floor muscles precedes rapid upper limb movements. 2002.
- [Result] Campos RM, Lucio AC, Lopes MHBM, Hacad CR, Perissinotto MCR, Glazer HI, D'Ancona CAL. Pelvic floor muscle training alone or in combination with oxybutynin in treatment of nonmonosymptomatic enuresis. A randomized controlled trial with 2-year follow up. Einstein (Sao Paulo). 2019 Jun 27;17(3):eAO4602. doi: 10.31744/einstein_journal/2019AO4602. PMID 31271608
- [Result] Ma Y, Liu X, Shen Y. Effect of traditional Chinese and Western medicine on nocturnal enuresis in children and indicators of treatment success: Randomized controlled trial. Pediatr Int. 2017 Nov;59(11):1183-1188. doi: 10.1111/ped.13417. PMID 28891253
- [Result] Vesna ZD, Milica L, Stankovic I, Marina V, Andjelka S. The evaluation of combined standard urotherapy, abdominal and pelvic floor retraining in children with dysfunctional voiding. J Pediatr Urol. 2011 Jun;7(3):336-41. doi: 10.1016/j.jpurol.2011.02.028. Epub 2011 Apr 27. PMID 21527231
- [Result] Hamano S, Yamanishi T, Igarashi T, Ito H, Murakami S. Functional bladder capacity as predictor of response to desmopressin and retention control training in monosymptomatic nocturnal enuresis. Eur Urol. 2000 Jun;37(6):718-22. doi: 10.1159/000020224. PMID 10828674
- [Result] Shah, V., T. PalEkar, and P. GuruPraSad, Surface Electromyography of Perianal Muscles in Children with and without Enuresis: A Cross-sectional Study. JOURNAL OF CLINICAL AND DIAGNOSTIC RESEARCH, 2022. 16(1): p. SC01-SC03.
- [Result] Abd El-Moghny, S.M., et al., Pelvic Floor Muscles Activity Deviation from the Normal among Children with Primary Monosymptomatic Nocturnal Enuresis. 2019.
- [Result] Haid B, Tekgul S. Primary and Secondary Enuresis: Pathophysiology, Diagnosis, and Treatment. Eur Urol Focus. 2017 Apr;3(2-3):198-206. doi: 10.1016/j.euf.2017.08.010. Epub 2017 Sep 6. PMID 28888814
- [Result] Neveus T. Pathogenesis of enuresis: Towards a new understanding. Int J Urol. 2017 Mar;24(3):174-182. doi: 10.1111/iju.13310. Epub 2017 Feb 16. PMID 28208214
- [Result] Kawauchi A, Tanaka Y, Naito Y, Yamao Y, Ukimura O, Yoneda K, Mizutani Y, Miki T. Bladder capacity at the time of enuresis. Urology. 2003 May;61(5):1016-8. doi: 10.1016/s0090-4295(02)02515-3. PMID 12736027
- [Result] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Walle JV, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: Update report from the standardization committee of the International Children's Continence Society. Neurourol Urodyn. 2016 Apr;35(4):471-81. doi: 10.1002/nau.22751. Epub 2015 Mar 14. PMID 25772695